CLINICAL TRIAL: NCT00001259
Title: The Treatment of Menstrually-Related Mood Disorders With the Gonadotropin Releasing Hormone (GnRH) Agonist, Depot Leuprolide Acetate (Lupron)
Brief Title: A Treatment Study for Premenstrual Syndrome (PMS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 900088; 90-M-0088
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2021-01-04

CONDITIONS: Premenstrual Syndrome; Menstruation Disturbances
Keywords: Depression; Menstrual Cycle; Gonadal Steroids; Estradiol; Progesterone; Mood Disorders
MeSH Terms: conditions — Premenstrual Syndrome; Menstruation Disturbances; Depression; Mood Disorders | interventions — Leuprolide; Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Study 1, Phase 1, Assignment 1 - Placebo (Placebo Comparator): As part of double Blind randomized trial, participants in Assignment 1 were randomized to 8 weeks of placebo (P) injections (1 injection per month). These participants then continued on to Study 2 after completion of 8 weeks of placebo injections.
  Interventions: Drug: Placebo injection
- Study 1, Phase 1, Assignment 2 - GnRH agonist injections (Lupron-L only) (Experimental): As part of double Blind randomized trial, participants in Assignment 2 were randomized to 8 weeks of GnRH agonist treatment 3.75 mg given intramuscularly monthly. Those who exhibited a remission of symptoms after 8 weeks continued on to receive one more month of GnRH agonist treatment (12 weeks total) and then entered Study 1, Phase 2.
  Interventions: Drug: Leuprolide
- Study 1, Phase 2, Arm 1 - Estradiol, then progesterone (Experimental): 12 weeks of GnRH agonist treatment 3.75 mg given intramuscularly monthly. Additionally, 4 weeks of transdermal Estradiol (100mcg/day by skin patch) and placebo suppositories. Week 5 involves 100mcg/day transdermal Estradiol and active Progesterone suppositories (200mg vaginally twice/day). Followed by 1-2 weeks (weeks 6-7) washout period. Then crossover to 5 weeks (week 8-12) of Progesterone suppositories (200mg vaginally twice/day) and placebo patches.
  Interventions: Drug: Leuprolide; Drug: Estradiol Patches; Drug: Progesterone; Drug: Placebo patch; Drug: Placebo suppository
- Study 1, Phase 2, Arm 2 - Progesterone, then estradiol (Experimental): 12 weeks of GnRH agonist treatment 3.75 mg given intramuscularly monthly. Additionally, 5 weeks of Progesterone suppositories (200mg vaginally twice/day) and placebo patches. Followed by 1-2 weeks (weeks 6-7) washout period. Then crossover to 4 weeks (weeks 8-11) of transdermal Estradiol (100mcg/day by skin patch) and placebo suppositories. Week 12 involves 100mcg/day transdermal Estradiol and active Progesterone suppositories (200mg vaginally twice/day).
  Interventions: Drug: Leuprolide; Drug: Estradiol Patches; Drug: Progesterone; Drug: Placebo patch; Drug: Placebo suppository
- Study 2, Phase 1 - GnRH agonist injections (Lupron-L only) (Experimental): Eight to 12 weeks of GnRH agonist treatment 3.75 mg given intramuscularly monthly.
  Interventions: Drug: Leuprolide
- Study 2, Phase 2, Arm 1 - Estradiol, then progesterone (Experimental): 12 weeks of GnRH agonist treatment 3.75 mg given intramuscularly monthly. Additionally, 4 weeks of transdermal Estradiol (100mcg/day by skin patch) and placebo suppositories. Week 5 involves 100mcg/day transdermal Estradiol and active Progesterone suppositories (200mg vaginally twice/day). Followed by 1-2 weeks (weeks 6-7) washout period. Then crossover to 5 weeks (week 8-12) of Progesterone suppositories (200mg vaginally twice/day) and placebo patches.
  Interventions: Drug: Leuprolide; Drug: Estradiol Patches; Drug: Progesterone; Drug: Placebo patch; Drug: Placebo suppository
- Study 2, Phase 2, Arm 2 - Progesterone, then estradiol (Experimental): 12 weeks of GnRH agonist treatment 3.75 mg given intramuscularly monthly. Additionally, 5 weeks of Progesterone suppositories (200mg vaginally twice/day) and placebo patches. Followed by 1-2 weeks (weeks 6-7) washout period. Then crossover to 4 weeks (weeks 8-11) of transdermal Estradiol (100mcg/day by skin patch) and placebo suppositories. Week 12 involves 100mcg/day transdermal Estradiol and active Progesterone suppositories (200mg vaginally twice/day).
  Interventions: Drug: Leuprolide; Drug: Estradiol Patches; Drug: Progesterone; Drug: Placebo patch; Drug: Placebo suppository

INTERVENTIONS:
Drug: Leuprolide — Eight to 12 weeks of GnRH agonist, Leuprolide Acetate 3.75 mg given intramuscularly monthly
  Arms: Study 1, Phase 1, Assignment 2 - GnRH agonist injections (Lupron-L only); Study 1, Phase 2, Arm 1 - Estradiol, then progesterone; Study 1, Phase 2, Arm 2 - Progesterone, then estradiol; Study 2, Phase 1 - GnRH agonist injections (Lupron-L only); Study 2, Phase 2, Arm 1 - Estradiol, then progesterone; Study 2, Phase 2, Arm 2 - Progesterone, then estradiol
Drug: Estradiol Patches — Transdermal Estradiol, 100mcg/day by skin patch
  Arms: Study 1, Phase 2, Arm 1 - Estradiol, then progesterone; Study 1, Phase 2, Arm 2 - Progesterone, then estradiol; Study 2, Phase 2, Arm 1 - Estradiol, then progesterone; Study 2, Phase 2, Arm 2 - Progesterone, then estradiol
Drug: Progesterone — Progesterone suppository, 200mg vaginally twice/day
  Arms: Study 1, Phase 2, Arm 1 - Estradiol, then progesterone; Study 1, Phase 2, Arm 2 - Progesterone, then estradiol; Study 2, Phase 2, Arm 1 - Estradiol, then progesterone; Study 2, Phase 2, Arm 2 - Progesterone, then estradiol
Drug: Placebo patch — Placebo by skin patch
  Arms: Study 1, Phase 2, Arm 1 - Estradiol, then progesterone; Study 1, Phase 2, Arm 2 - Progesterone, then estradiol; Study 2, Phase 2, Arm 1 - Estradiol, then progesterone; Study 2, Phase 2, Arm 2 - Progesterone, then estradiol
Drug: Placebo injection — Placebo given intramuscularly monthly
  Arms: Study 1, Phase 1, Assignment 1 - Placebo
Drug: Placebo suppository — Placebo vaginal suppository
  Arms: Study 1, Phase 2, Arm 1 - Estradiol, then progesterone; Study 1, Phase 2, Arm 2 - Progesterone, then estradiol; Study 2, Phase 2, Arm 1 - Estradiol, then progesterone; Study 2, Phase 2, Arm 2 - Progesterone, then estradiol

SUMMARY:
This study examines the effects of estrogen and progesterone on mood, the stress response, and brain function and behavior in women with premenstrual syndrome.

Previously this study has demonstrated leuprolide acetate (Lupron (Registered Trademark)) to be an effective treatment for PMS. The current purpose of this study is to evaluate how low levels of estrogen and progesterone (that occur during treatment with leuprolide acetate) compare to menstrual cycle levels of estrogen and progesterone (given during individual months of hormone add-back) on a variety of physiologic measures (brain imaging, stress testing, etc.) in women with PMS.

PMS is a condition characterized by changes in mood and behavior that occur during the second phase of the normal menstrual cycle (luteal phase). This study will investigate possible hormonal causes of PMS by temporarily stopping the menstrual cycle with leuprolide acetate and then giving, in sequence, the menstrual cycle hormones progesterone and estrogen. The results of these hormonal studies will be compared between women with PMS and healthy volunteers without PMS (see also protocol 92-M-0174).

At study entry, participants will undergo a physical examination. Blood, urine, and pregnancy tests will be performed. Cognitive functioning and stress response will be evaluated during the study along with brain imaging and genetic studies.

DETAILED DESCRIPTION:
This protocol is designed to accompany Clinical Protocol # 81-M-0126, The Phenomenology and Biophysiology of Menstrually-Related Mood and Behavioral Disorders. Its original purposes were as follows: 1) to evaluate the efficacy of the gonadotropin releasing hormone (GnRH) agonist depot leuprolide acetate (Lupron) in the treatment of menstrually-related mood disorders (MRMD) by determining whether mood and behavioral symptoms are eliminated when the cyclic secretion of both gonadotropic hormones and gonadal steroids is suppressed, and 2) to determine the possible relevance of gonadal steroids to affective state by sequentially replacing estradiol and progesterone during continued GnRH suppression in those patients whose premenstrual symptoms remit following administration of the GnRH agonist. We observed that GnRH agonist induced ovarian suppression was an effective treatment compared to placebo in women with MRMD. Additionally, women with MRMD but not asymptomatic controls (participating in companion protocol 92-M-0174) experienced a recurrence of mood and behavioral symptoms when either estradiol or progesterone (but not placebo) was added back. These data suggest that women with MRMD have a differential sensitivity to the mood destabilizing effects of gonadal steroids.

Having established that women with MRMD show a differential behavioral response to estrogen and progesterone, we now hope to identify the underlying mechanisms and physiologic concomitants of the differential behavioral sensitivity by performing studies (described in companion protocols) under the three hormonal conditions created by this protocol, and comparing results obtained with those seen in normal controls (Protocol #92-M-0174). Planned studies include the following: cognitive testing, brain imaging [(3D-positron emission tomography (PET), functional magnetic resonance imaging (FMRI), magnetic resonance spectroscopy (MRS)] and genetic studies including induced pluripotent cells.

ELIGIBILITY:
* INCLUSION CRITERIA:

The subjects of this study will be women who meet the criteria for MRMD as described in Protocol No. 81-M-0126, 'The Phenomenology and Biophysiology of Menstrually-related Mood and Behavioral Disorders.' In brief, these criteria include:

1. history within the last two years of at least six months with menstrually-related mood or behavioral disturbances of at least moderate severity--i.e., disturbances that are distinct in appearance and associated with a notable degree of subjective distress;
2. symptoms should have a sudden onset and offset;
3. age 18-50;
4. not pregnant and in good medical health;
5. medication free.

   All patients participating in this protocol will have already participated in Protocol No. 81-M-0126 and will have a prospectively confirmed and predictable relationship between their mood disorder and the premenstrual phase of the menstrual cycle, i.e., a 30% change in severity of symptom self rating scales, relative to the range of the scale employed, during the seven days premenstrually compared with the seven days post-menstrually in two out of three months of study.

   The Schedule for Affective Disorders and Schizophrenia will be administered to all patients prior to study entry. Any patient with a current axis I psychiatric diagnosis will be excluded from participating in this protocol.

   Prior to treatment, a complete physical and neurological examination will have been performed and the following routine laboratory data obtained:

   A. Blood

   Complete blood count; thyroid function tests; cortisol; renal function tests, such as blood urea nitrogen (BUN) and creatinine; electrolytes; glucose; liver function tests.

   B. Urine

   Routine urinalysis; urine pregnancy test.

   GnRH agonist will not be administered to any subject with significant clinical or laboratory abnormalities. The blood tests and urinalysis will be repeated 2 weeks after GnRH agonist administration to rule out any evidence of acute renal, hepatic or hematologic toxicity.

   Results of Pap smear performed within one year of the onset of treatment will be obtained.

   EXCLUSION CRITERIA:

   The following conditions will constitute contraindications to treatment with hormonal therapy and will preclude a subject's participation in this protocol:
   * current Axis I psychiatric diagnosis
   * history consistent with endometriosis,
   * diagnosis of ill-defined, obscure pelvic lesions, particularly, undiagnosed ovarian enlargement,
   * hepatic disease as manifested by abnormal liver function tests,
   * history of mammary carcinoma,
   * history of pulmonary embolism or phlebothrombosis
   * undiagnosed vaginal bleeding
   * porphyria
   * diabetes mellitus
   * history of malignant melanoma
   * cholecystitis or pancreatitis,
   * cardiovascular or renal disease
   * pregnancy
   * Any woman meeting the Stages of Reproductive Aging Workshop Criteria (STRAW) for the perimenopause. Specifically, we will exclude any woman with an elevated plasma follicle stimulating hormone (FSH) level (>= 14 IU/L) and with menstrual cycle variability of > 7 days different from their normal cycle length.
   * Subjects taking birth control pills will be excluded from the study.
   * Subjects taking diuretics, prostaglandin inhibitors, or pyridoxine (putative treatments for MRMD) will similarly be excluded from the study
   * Patients taking psychotropic agents (e.g., lithium carbonate, tricyclic antidepressants).
   * All subjects will be required to use non-hormonal forms of birth control (e.g., barrier methods) to avoid pregnancy during this study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 1992-08-11 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Schmidt, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rubinow DR, Hoban MC, Grover GN, Galloway DS, Roy-Byrne P, Andersen R, Merriam GR. Changes in plasma hormones across the menstrual cycle in patients with menstrually related mood disorder and in control subjects. Am J Obstet Gynecol. 1988 Jan;158(1):5-11. doi: 10.1016/0002-9378(88)90765-x. PMID 2962499
- [Background] Schmidt PJ, Nieman LK, Grover GN, Muller KL, Merriam GR, Rubinow DR. Lack of effect of induced menses on symptoms in women with premenstrual syndrome. N Engl J Med. 1991 Apr 25;324(17):1174-9. doi: 10.1056/NEJM199104253241705. PMID 2011161
- [Background] Schmidt PJ, Nieman LK, Danaceau MA, Adams LF, Rubinow DR. Differential behavioral effects of gonadal steroids in women with and in those without premenstrual syndrome. N Engl J Med. 1998 Jan 22;338(4):209-16. doi: 10.1056/NEJM199801223380401. PMID 9435325
- [Derived] Li HJ, Goff A, Rudzinskas SA, Jung Y, Dubey N, Hoffman J, Hipolito D, Mazzu M, Rubinow DR, Schmidt PJ, Goldman D. Altered estradiol-dependent cellular Ca2+ homeostasis and endoplasmic reticulum stress response in Premenstrual Dysphoric Disorder. Mol Psychiatry. 2021 Nov;26(11):6963-6974. doi: 10.1038/s41380-021-01144-8. Epub 2021 May 25. PMID 34035477
- [Derived] Di Florio A, Alexander D, Schmidt PJ, Rubinow DR. Progesterone and plasma metabolites in women with and in those without premenstrual dysphoric disorder. Depress Anxiety. 2018 Dec;35(12):1168-1177. doi: 10.1002/da.22827. Epub 2018 Sep 5. PMID 30184299
- [Derived] Nguyen TV, Reuter JM, Gaikwad NW, Rotroff DM, Kucera HR, Motsinger-Reif A, Smith CP, Nieman LK, Rubinow DR, Kaddurah-Daouk R, Schmidt PJ. The steroid metabolome in women with premenstrual dysphoric disorder during GnRH agonist-induced ovarian suppression: effects of estradiol and progesterone addback. Transl Psychiatry. 2017 Aug 8;7(8):e1193. doi: 10.1038/tp.2017.146. PMID 28786978
- [Derived] Dubey N, Hoffman JF, Schuebel K, Yuan Q, Martinez PE, Nieman LK, Rubinow DR, Schmidt PJ, Goldman D. The ESC/E(Z) complex, an effector of response to ovarian steroids, manifests an intrinsic difference in cells from women with premenstrual dysphoric disorder. Mol Psychiatry. 2017 Aug;22(8):1172-1184. doi: 10.1038/mp.2016.229. Epub 2017 Jan 3. PMID 28044059
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1990-M-0088.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant signed consent but withdrew prior to study start
Pre-assignment Details: 8 of 46 participants who completed Study 2, Phase 1 did not proceed to Study 2, Phase 2.
Period: Study 1
Arm/Group | Study 1, Phase 1, Assignment 1 - Placebo | Study 1, Phase 1, Assignment 2 - GnRH Agonist Injections (Lupron-L Only) | Study 1, Phase 2, Arm 1 - Estradiol, Then Progesterone | Study 1, Phase 2, Arm 2 - Progesterone, Then Estradiol | Study 2, Phase 1 - GnRH Agonist Injections (Lupron-L Only) | Study 2, Phase 2, Arm 1 - Estradiol, Then Progesterone | Study 2, Phase 2, Arm 2 - Progesterone, Then Estradiol
Started | 10 | 10 | 0 | 0 | 0 | 0 | 0
Completed Phase 1 | 10 | 10 | 0 | 0 | 0 | 0 | 0
Started Phase 2 | 0 | 0 | 4 (4 of 10 participants from Study 1, Phase 1, Assignment 2 - GnRH agonist injections (Lupron-L only) were randomized to this arm) | 6 (6 of 10 participants from Study 1, Phase 1, Assignment 2 - GnRH agonist injections (Lupron-L only) were randomized to this arm) | 0 | 0 | 0
Completed Phase 2 | 0 | 0 | 4 | 5 (one participant dropped off due to adverse reaction) | 0 | 0 | 0
Started Phase 2 - Crossover Arm | 0 | 0 | 4 | 5 | 0 | 0 | 0
Completed Phase 2 - Crossover Arm | 0 | 0 | 4 | 5 | 0 | 0 | 0
Completed | 10 | 10 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Study 2
Arm/Group | Study 1, Phase 1, Assignment 1 - Placebo | Study 1, Phase 1, Assignment 2 - GnRH Agonist Injections (Lupron-L Only) | Study 1, Phase 2, Arm 1 - Estradiol, Then Progesterone | Study 1, Phase 2, Arm 2 - Progesterone, Then Estradiol | Study 2, Phase 1 - GnRH Agonist Injections (Lupron-L Only) | Study 2, Phase 2, Arm 1 - Estradiol, Then Progesterone | Study 2, Phase 2, Arm 2 - Progesterone, Then Estradiol
Started | 0 | 0 | 0 | 0 | 48 (Include 9 subjects from Study 1, Phase 1, Assignment 1 - Placebo) | 0 | 0
Completed Phase 1 | 0 | 0 | 0 | 0 | 46 | 0 | 0
Started Phase 2 | 0 | 0 | 0 | 0 | 0 | 21 | 17
Completed Phase 2 | 0 | 0 | 0 | 0 | 0 | 21 | 17
Started Phase 2 - Crossover Arm | 0 | 0 | 0 | 0 | 0 | 21 | 17
Completed Phase 2 - Crossover Arm | 0 | 0 | 0 | 0 | 0 | 21 | 17
Completed | 0 | 0 | 0 | 0 | 46 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants either received placebo or GnRH agonist injections (Lupron-L only) prior to randomization to any arm in either study.
Groups:
- Placebo: 8 weeks of placebo (P) injections (one injection per month)
- GnRH Agonist Injections (Lupron-L Only): Eight to 12 weeks of GnRH agonist treatment 3.75 mg given intramuscularly monthly before randomization to estradiol or progesterone arm in the crossover phase of the study
- Total: Total of all reporting groups
Arm/Group | Placebo | GnRH Agonist Injections (Lupron-L Only) | Total
Number analyzed (Participants) | 10 | 49 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 49 | 59
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 49 | 59
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 10 | 47 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 15 | 15
  White | 10 | 29 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Beck Depression Inventory Score
Description: The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures the severity of symptoms accompanying depression. Each item has a minimum score of 0 and a maximum score of 3, with higher numbers consistent with more severe symptoms. The score of each item is summed to amount the overall BDI score, with a minimum score of 0 and a maximum score of 63. Higher BDI scores are consistent with more severe depression. Score of 16 or greater is consistent with clinical depression.
  Each participant completed the BDI every 2 weeks during each of the study phases throughout the 6-month study. Outcome measures reported consist of the average of two BDI scores from each phase of the study: the last 4 weeks of the GnRH agonist alone; weeks 6 and 8 of placebo alone; during the 4-week long estradiol phase (weeks 2 and 4 of estradiol) and the 4-week long progesterone phase (weeks 2 and 4 of progesterone).
Time Frame: Placebo: Weeks 6 and 8 of Placebo; Lupron only: Weeks 6 and 8 or 10 and 12; Estradiol or progesterone: Weeks 2 and 4
Population: Analyses included comparison of participants mean BDI scores during each phase of the study
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Estradiol: 4 weeks of transdermal Estradiol (100mcg/day by skin patch)
- Progesterone: 5 weeks of Progesterone suppositories (200mg vaginally twice/day)
Arm/Group | Placebo | GnRH Agonist Injections (Lupron-L Only) | Estradiol | Progesterone
Number analyzed (Participants) | 10 | 48 | 48 | 48
score on a scale | 2.6 (2.6) | 3.0 (3.8) | 5.3 (5.3) | 3.6 (5.7)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Placebo | GnRH Agonist Injections (Lupron-L Only) | Estradiol | Progesterone
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/58 | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/58 | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/10 | 2/58 | 3/48 | 0/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | GnRH Agonist Injections (Lupron-L Only) (N=58) | Estradiol (N=48) | Progesterone (N=48)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital atrophy (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/59/NCT00001259/Prot_SAP_000.pdf